CLINICAL TRIAL: NCT01888315
Title: Safety and Efficacy Study Investigating the Effects of Catheter-based Renal Denervation on Different Organ Systems in Patients With Increased Sympathetic Activity
Brief Title: Influence of Catheter-based Renal Denervation in Diseases With Increased Sympathetic Activity
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Symplicity Extension
Record Dates: First submitted 2012-09-04; First posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Hypertension; Heart Failure; Chronic Kidney Disease; Diabetes; Heart Rhythm Disorders
Keywords: Hypertension; Heart Failure; Sympathetic activity
MeSH Terms: conditions — Hypertension; Heart Failure; Renal Insufficiency, Chronic; Diabetes Mellitus; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Catheter-based renal denervation (Experimental): One procedure will be performed using one of the CE-marked devices for renal denervation:
  Device: Renal denervation with Symplicity Flex Medtronic/Ardian Device: Renal denervation with EnligHTN St. Jude Medical Device: Renal denervation with Paradise Recor Device: Renal denervation with V2 Vessix
  Interventions: Device: Renal denervation with Symplicity Flex Medtronic/Ardian; Device: Renal denervation with EnligHTN St. Jude Medical; Device: Renal denervation with Paradise Recor; Device: Renal denervation with V2 Vessix
- Medical therapy (No Intervention): Best medical therapy using guideline recommended drugs in each disease state.

INTERVENTIONS:
Device: Renal denervation with Symplicity Flex Medtronic/Ardian — Renal denervation using CE-marked devices will be performed according to best medical practice.
  Arms: Catheter-based renal denervation
Device: Renal denervation with EnligHTN St. Jude Medical — Renal denervation using CE-marked devices will be performed according to best medical practice.
  Arms: Catheter-based renal denervation
Device: Renal denervation with Paradise Recor — Renal denervation using CE-marked devices will be performed according to best medical practice.
  Arms: Catheter-based renal denervation
Device: Renal denervation with V2 Vessix — Renal denervation using CE-marked devices will be performed according to best medical practice.
  Arms: Catheter-based renal denervation

SUMMARY:
The study is aiming to document the long-term safety and effectiveness of renal denervation in patients with hypertension and other diseases characterized by elevated sympathetic drive. Catheter-based renal denervation will be performed using CE marked, percutaneous, systems.

DETAILED DESCRIPTION:
Inclusion Criteria

1. Individual is 18 years of age.
2. Individual agrees to have all procedures performed, and is competent and willing to provide written, informed consent to participate in the registry.
3. Patient scheduled for renal sympathetic denervation using market-released device.

Exclusion Criteria

1. In the eyes of the treating physician, the renal artery anatomy would interfere with safe cannulation of the renal artery or meets local standards for surgical repair.
2. Individual has any serious medical condition, which in the opinion of the treating physician may adversely affect the safety and/or effectiveness of the participant (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, hemophilia, significant anemia, etc.).

ELIGIBILITY:
Inclusion Criteria

1. Individual is 18 years of age.
2. Individual agrees to have all procedures performed, and is competent and willing to provide written, informed consent to participate in the registry.
3. Patient scheduled for renal sympathetic denervation using market-released device.

Exclusion Criteria

1. In the eyes of the treating physician, the renal artery anatomy would interfere with safe cannulation of the renal artery or meets local standards for surgical repair.
2. Individual has any serious medical condition, which in the opinion of the treating physician may adversely affect the safety and/or effectiveness of the participant (i.e., patients with clinically significant peripheral vascular disease, abdominal aortic aneurysm, bleeding disorders such as thrombocytopenia, hemophilia, significant anemia, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2011-01; Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of renal denervation | Baseline to 6 months
  Effect on blood pressure including office, ABPM, and home-based measurements.
  Number of adverse events (death, stroke, myocardial infarction, new dialysis, and congestive heart failure).
  Changes of antihypertensive medications.
  Effects on renal function assessed with glomerular filtration rate.
  Renovascular safety (renal artery stenosis) assessed by duplex ultrasound.

SECONDARY OUTCOMES:
Effect of renal denervation on different organ systems. | Baseline, 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Myocardial function and geometry using echo and MRI.
  Heart rate changes and arrhythmias.
  Glucose metabolism and insulin resistance (fasting and during oGTT).
  Hospitalization rates (eg. hypertensive emergencies, heart failure, etc).
Safety and efficacy of renal denervation | Baseline, 3, 12, 18, 24, 30, 36, 42, 48, 54, 60 months
  Effect on blood pressure including office, ABPM, and home-based measurements.
  Number of adverse events (death, stroke, myocardial infarction, new dialysis, and congestive heart failure).
  Changes of antihypertensive medications.
  Effects on renal function assessed with glomerular filtration rate.
  Renovascular safety (renal artery stenosis) assessed by duplex ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Felix Mahfoud, MD, Study Director — University Hospital, Saarland; Michael Böhm, MD, Principal Investigator — University Hospital, Saarland
Locations (1):
- University Hospital Saarland, Homburg/Saar, Germany

REFERENCES:
- [Derived] Lauder L, Siwy J, Mavrogeorgis E, Keller F, Kunz M, Wachter A, Emrich IE, Bohm M, Mischak H, Mahfoud F. Impact of Renal Denervation on Urinary Peptide-Based Biomarkers in Hypertension. Hypertension. 2024 Jun;81(6):1374-1382. doi: 10.1161/HYPERTENSIONAHA.124.22819. Epub 2024 Apr 4. PMID 38572643